CLINICAL TRIAL: NCT01404936
Title: A Phase II Study of a-Interferon With Adriamycin, Bleomycin, Velban, and Dacarbazine (ABVD) for Patients With Hodgkin's Disease
Brief Title: Study of a-Interferon With Adriamycin, Bleomycin, Velban, and Dacarbazine (ABVD) With Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM96-060
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Results first posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: Lymphoma; Hodgkin's Disease; Stage III and IV; Adriamycin; Doxorubicin; Rubex; Bleomycin; Bleomycin Sulfate; BLM; Dacarbazine; DTIC-DOME; Interferon-2A; Interferon-Alfa-2a; Roferon-A; Velban; Vinblastine
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Interferon alpha-2; Doxorubicin; Bleomycin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon-2A + Chemotherapy (Experimental): Interferon-2A 4 (x106 IU/m^2) subcutaneously Day 1 - 4 + ABVD Chemotherapy on Day 4 (ABVD: Adriamycin 25 mg/m2 intravenous (IV), Bleomycin 10 mg/m^2 IV, Velban 6 mg/m2 IV, and Dacarbazine 375 mg/m2 IV)
  Interventions: Drug: Interferon-2A; Drug: Adriamycin; Drug: Bleomycin; Drug: Velban; Drug: Dacarbazine

INTERVENTIONS:
Drug: Interferon-2A — 4 (x106 IU/m^2) subcutaneously on days 1-4.
  Other Names: Interferon-Alfa-2a; Roferon-A
Drug: Adriamycin — 25 mg/m^2 by vein on day 4.
  Other Names: Doxorubicin; Rubex
Drug: Bleomycin — 10 mg/m^2 by vein on day 4.
  Other Names: Bleomycin Sulfate; BLM
Drug: Velban — 6 mg/m^2 by vein on day 4.
  Other Names: Vinblastine
Drug: Dacarbazine — 375 mg/m^2 by vein on day 4.
  Other Names: DTIC-DOME

SUMMARY:
This is a clinical research study of interferon (IFN) plus chemotherapy with the standard combination of Adriamycin, Bleomycin, Velban, and Dacarbazine (ABVD). The treatment will be given to patients with Hodgkin's disease. The study will look at whether adding IFN to ABVD improves the immune response against Hodgkin's disease, and will determine whether the toxicity of ABVD is increased by adding IFN.

DETAILED DESCRIPTION:
Each treatment cycle will last 2 weeks. On days 1 - 4 of each cycle, patients will be given a shot of IFN under the skin. On day 4, patients will be given ABVD through a vein over one-hour.

The plan is for patients to receive 12 cycles of treatment. However, patients will leave the study if they have severe side effects or if the cancer grows or spreads. They will also leave if the cancer does not improve after 6 cycles. Patient who leave the study will be offered other treatments. A maximum of 35 patients will be treated with that dose.

Before the first treatment, patient will have a physical exam, blood tests, and a heart scan. Within 1 month of starting treatment, patients will have a chest X-ray, CT scans of the abdomen and pelvis, and a gallium scan.

During the study, patient will have blood tests every week and a physical exam every 2 weeks. The X-ray, CT scans, and gallium scan will be repeated after cycles 6 and 12.

All the drugs in this study are approved by the U.S. Food and Drug Administration and are available by prescription. ABVD is a standard treatment for Hodgkin's disease; IFN is an investigational treatment for Hodgkin's disease. About 35 patients will be enrolled in the study. All treatment will be given in the outpatient clinic at M.D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Hodgkin's disease patients who relapse after radiation therapy alone, or in combination with Novantrone, Oncovin, Velban, and Prednisone (NOVP); and previously untreated patients with stage III and IV who are eligible for standard ABVD therapy.
2. Must have adequate bone marrow reserve Absolute neutrophil count (ANC) > 1,000/uL, Platelets > 100,000
3. Left ventricular ejection fraction (LVEF) >/= 50%, serum creatinine < 2mg/dl, serum bilirubin < 2mg/dl

Exclusion Criteria:

1. No prior therapy with Mustargen Oncovin Procarbazine Prednisone (MOPP).
2. No severe pulmonary disease including Chronic obstructive pulmonary disease (COPD) and asthma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1996-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 25, 1996 through March 3, 2000. All participants were recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 35 participants registered, five (5) were excluded from the trial.
Period: Overall Study
Arm/Group | Interferon-2A + Chemotherapy
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interferon-2A + Chemotherapy
Number analyzed (Participants) | 30
Age Continuous [Median (Full Range); unit: years] | 30 [18 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Participants' Response
Description: Complete Response (CR): Disappearance of all clinical evidence of active tumors for a minimum of 8 weeks. Partial Response (PR): 50% or greater decrease in sum of products all measured lesions persisting for at least 4 weeks. No Change: Steady state or change of +/- 25% of tumor size and no progression for minimum of 8 weeks with no appearance of new lesions. Progressive Disease: > 25 % increase in size of any measurable lesion or appearance of significant new lesions.
Time Frame: After 6 courses (3 months)
Population: Two patients did not complete therapy; however, they were included in the intent-to-treat analysis. One patient was censored at the last follow-up date since no events had occurred.
Measure: Number; unit: participants
Arm/Group | Interferon-2A + Chemotherapy
Number analyzed (Participants) | 30
participants
  Complete Response | 23
  Uncomfirmed Complete Response | 2
  Partial Response | 3
  Progressive Disease | 1

ADVERSE EVENTS:
Time Frame: 3 years and 4 months
Arm/Group | Interferon-2A + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon-2A + Chemotherapy (N=30)
Cytopenia (Blood and lymphatic system disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon-2A + Chemotherapy (N=30)
Asthenia (General disorders) | 2
Fever (Investigations) | 10
Nausea (Gastrointestinal disorders) | 20
Psychiatric Disorders (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No